CLINICAL TRIAL: NCT06079021
Title: COOLEY- Study: ACute on ChrOnic Liver FailurE Using the CYtosorb Device
Acronym: COOLEY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: CytoSorbents Europe GmbH (Industry)
Responsible Party: Principal Investigator, Karolien Dams, Principal Investigator, MD, senior staff intensive care, University Hospital, Antwerp
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Edge 2930
Record Dates: First submitted 2023-07-26; First posted 2023-10-12 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Acute-On-Chronic Liver Failure; Anticoagulant Adverse Reaction; Sarcopenia; Ultrasonography
Keywords: acute on chronic liver failure; sarcopenia; citrate anticoagulation; low molecular weight heparins; hand grip strength; skeletal muscle ultrasound; hemoadsorption; CRRT
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Application of CytoSorb treatment to ACLF patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CytoSorb hemoadsorption (Active Comparator): Patients with acute on chronic liver failure will receive CytoSorb treatment for 72 hours. The aim is to remove the molecules that drive systemic inflammation.
  Interventions: Device: CytoSorb
- Control group (No Intervention): Historical group that received only standard medical care

INTERVENTIONS:
Device: CytoSorb — Application of CytoSorb treatment for 72 hours in patients with ACLF
  Arms: CytoSorb hemoadsorption

SUMMARY:
A Prospective, Single-Center trial, in Patients With Acute on Chronic Liver Failure. Study of Standard Medical Care Plus CytoSorb® Compared to Standard Medical Care Alone in a historical group.

DETAILED DESCRIPTION:
The study team wants to investigate the effect of Cytosorb hemoadsorption on the bilirubin level as well as on the ammonia level changes induced by the therapy in patients with Acute on Chronic Liver Failure (ACLF) .

In this group of patients with ACLF grade 2 and 3 the investigators want to determine the prevalence and development of sarcopenia by sequential quadriceps and thenar ultrasound images and by handgrip strength measurement.

The investigators will objectify muscle mass by skeletal muscle ultrasound of quadriceps and thenar muscles in this sickest subgroup of cirrhotic patients. Ultrasound forms a part of the daily clinical routine in ICU. The study team wants to compare both measurements and objectify the evolution to study the reliability and validity of ultrasound to quantify muscles in chronic liver disease and its clinical values. Most of ultrasonographic studies are based on quadriceps exploration, which is more inconvenient and takes more time than exploring the hands because patients need to remove clothes and lie down. The study team also hypothesizes that thenar muscles are less subject to fluid overload than the quadriceps muscles are.

When available, lumbar skeletal muscle indices will be compared by computed tomography or magnetic resonance imaging.

In this group of patients with ACLF, receiving Continuous Renal Replacement Therapy (CRRT) the appropriate choice of anticoagulant remains controversial. The objective of this study is to compare the efficacy and safety of regional citrate anticoagulation (RCA) and Low Molecular Weight Heparin (LMWH) in critically ill ACLF patients requiring CRRT. These two commercially available anticoagulation methods are used in daily practice in the ICU. The first 10 patients will receive anticoagulation with LMWH with monitoring of anti-Xa. The second cohort of patients will receive RCA.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥ 18 years) admitted to the University Hospital of Antwerp (UZA), Belgium.

  * Written informed consent from patient or if not possible due to encephalopathy (> grade 2): legal representative
  * acute-on-chronic liver failure (ACLF) grade ≥ 2:

    * Acute decompensation event (identifiable trigger)
    * Hepatic encephalopathy grade ≥ 2
    * Acute kidney injury (AKI) according to Kidney Disease: Improving Global Outcome (KDIGO) criteria stage 3 (≥ 3-fold increase of serum creatinine OR increase of serum creatinine to ≥ 4 mg/dl OR urine output ≤ 0.3 ml/kg/h for ≥ 24 hours OR anuria for ≥ 12 hours)
    * Serum bilirubin ≥ 10 mg/dl
    * Hemodynamic instability with vasopressor support (norepinephrine > 0.05 mcg/kg/min)

Exclusion Criteria:

* • known patient will against participation in the study or against the measures applied in the study

  * a decision made prior to inclusion to stop further treatment of the patient within the next 24 hours
  * no complete remission of malignancy including hepatocellular carcinoma within the past 12 months
  * ongoing intermittent or CRRT before study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The impact of CytoSorb on serum bilirubin removal | 24 and 72 hours
  20 participants with a serum bilirubin of ≥ 10 mg/dl will undergo CytoSorb for 72 hours
Changes in ammonia and severity of hepatic encephalopathy during treatment period | 24 and 72 hours
  The West Haven criteria are used for grading the severity of hepatic encephalopathy, which include 5 grades ranging from minimal (slightly impaired) to grade IV (comatose)

SECONDARY OUTCOMES:
changes in hemodynamic profile | 24 and 72 hours
  Change in hemodynamic profile (i.e. mean arterial pressure normalized to norepinephrine equivalents) during the 72-h study intervention.
Vasopressors | 24 and 72 hours
  Duration of vasopressor support in days
ACLF (Acute on Chronic Liver Failure) Grading | first week
  Assessment of ACLF grading (minimum 0 - maximum 3; higher score means a worse outcome) during the 72h intervention up to 1 week after diagnosis of ACLF
SOFA Score | 0, 72 and 168 hours
  Changes in Sequential Organ Failure Assessment (SOFA) (minimum 0-maximum 24; higher score means a worse outcome) score during the 72h study period and up to 1 week after.
scores | 15 days
  Changes in CLIF-C (Chronic Liver Failure Consortium)(minimu 0 - maximum 100; higher score means a worse outcome) score during the 72-h intervention, up to 15 days after diagnosis of ACLF
Ventilation | 0, 24 and 72 hours
  Duration of mechanical ventilation,
Cytokines | 0, 24 and 72 hours
  Changes in cytokines (IL-6, IL-8, IL-16, TNF (tumor necrosis factor)-alpha) value (pg/ml)
Mortality | 28, 60 and 90 days after enrolment
  Mortality at 28, 60 and 90 days after enrolment
Improvement of Renal function after application of CytoSorb | 7, 14, 21 and 90 days after enrolment
  Acute kidney injury (AKI) according to Kidney Disease: Improving Global Outcome (KDIGO) criteria stage 3 (≥ 3-fold increase of serum creatinine OR increase of serum creatinine to ≥ 4 mg/dl OR urine output ≤ 0.3 ml/kg/h for ≥ 24 hours OR anuria for ≥ 12 hours) will receive CytoSorb treatmetn. Serum creatinine will be measured at day 7, 14, 21 and 90 days
Cytosorb filter | up to 28 days after enrolment
  Adverse events attributable to CytoSorb up to 28 days after enrolment
Change in Bile acids | 72 hours after enrolment
  Bile acids after 72 hours
Sarcopenia | 0, 24 and 72 hours
  Prevalence and development of sarcopenia
Anticoagulation | 0, 24 and 72 hours
  Adverse events attributable to anticoagulation
SAPS II score | Day 0, Day 3, Day 7
  Simplified Acute Physiology Score II (SAPS II) (minimum 0 - maximum 163; higher score means a worse outcome) during the 72-h study intervention and up to 1 week after
Change in inflammatory values: lactate | Day 0, Day 1 and Day 3
  measurement of lactate (reference < 2 mmol/L)
Change in inflammatory values: procalcitonin | Day 0, Day 1 and Day 3
  measurement of procalcitonin (reference < 0.5 ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Karolien Dams, Principal Investigator — University Hospital, Antwerp
Locations (1):
- UZA, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wlodzimirow KA, Eslami S, Abu-Hanna A, Nieuwoudt M, Chamuleau RA. A systematic review on prognostic indicators of acute on chronic liver failure and their predictive value for mortality. Liver Int. 2013 Jan;33(1):40-52. doi: 10.1111/j.1478-3231.2012.02790.x. Epub 2012 Mar 19. PMID 22429562
- [Background] Popescu M, David C, Marcu A, Olita MR, Mihaila M, Tomescu D. Artificial Liver Support with CytoSorb and MARS in Liver Failure: A Retrospective Propensity Matched Analysis. J Clin Med. 2023 Mar 14;12(6):2258. doi: 10.3390/jcm12062258. PMID 36983259
- [Background] Buchard B, Boirie Y, Cassagnes L, Lamblin G, Coilly A, Abergel A. Assessment of Malnutrition, Sarcopenia and Frailty in Patients with Cirrhosis: Which Tools Should We Use in Clinical Practice? Nutrients. 2020 Jan 9;12(1):186. doi: 10.3390/nu12010186. PMID 31936597
- [Background] Lopes J, Grams ST, da Silva EF, de Medeiros LA, de Brito CMM, Yamaguti WP. Reference equations for handgrip strength: Normative values in young adult and middle-aged subjects. Clin Nutr. 2018 Jun;37(3):914-918. doi: 10.1016/j.clnu.2017.03.018. Epub 2017 Mar 24. PMID 28389120
- [Background] Jacobs R, Verbrugghe W, Dams K, Roelant E, Couttenye MM, Devroey D, Jorens P. Regional Citrate Anticoagulation in Continuous Renal Replacement Therapy: Is Metabolic Fear the Enemy of Logic? A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Life (Basel). 2023 May 17;13(5):1198. doi: 10.3390/life13051198. PMID 37240843